CLINICAL TRIAL: NCT05789030
Title: Treatment Strategies for IgG4-RD Patients With Superficial Organ Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgG4-RD, superficial organ
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Autoimmune Diseases
Keywords: Immunoglobulin G4-Related Disease; treatment strategies; iguratimod; leflunomide; relapse
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease; Recurrence | interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination; iguratimod; Leflunomide; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Patients are treated with Diprospan (1mL im) and then with iguratimod (25mg bid) for 12 months
  Interventions: Drug: Diprospan plus iguratimod
- Group II (Experimental): Patients are treated with Diprospan (1mL im) and then with leflunomide (10-20mg qd) for 12 months.
  Interventions: Drug: Diprospan plus leflunomide
- Group Ⅲ (Experimental): Patients are treated with prednisone (20 mg qd and taper to ≦ 5mg in 3 months) and leflunomide (10-20mg qd) for 12 months.
  Interventions: Drug: Prednisone plus leflunomide

INTERVENTIONS:
Drug: Diprospan plus iguratimod — Patients are treated with Diprospan (1mL im) and then with iguratimod (25mg bid) for 12 months.
  Arms: Group I
Drug: Diprospan plus leflunomide — Patients are treated with Diprospan (1mL im) and then with leflunomide (10-20mg qd) for 12 months.
  Arms: Group II
Drug: Prednisone plus leflunomide — Patients are treated with prednisone (20 mg qd and taper to ≦ 5mg in 3 months) and leflunomide (10-20mg qd) for 12 months.
  Arms: Group Ⅲ

SUMMARY:
This study has been designed as a 12-month, open-label randomized controlled clinical trial. The study aims to compare the efficacy and safety of three treatment strategies in IgG4-RD patients with superficial organ involvement: Diprospan plus iguratimod, Diprospan plus leflunomide and prednisone plus leflunomide.

DETAILED DESCRIPTION:
90 IgG4-RD patients with superficial organ involvement are enrolled in this study and randomly divided into three groups at a 1:1:1 ratio: patients in group I are treated with Diprospan (1mL im) and then with iguratimod (25mg bid); patients in group Ⅱ are treated with Diprospan (1mL im) and then with leflunomide (10-20mg qd); and patients in group Ⅲ are treated with prednisone (20 mg qd and taper to ≦ 5mg in 3 months) and leflunomide (10-20mg qd). All patients will be followed up for 12 months, and clinical evaluations, laboratory tests, image examinations and IgG4-RD responder index (RI) will be recorded during follow up. The primary endpoint is the difference of relapse rate between two groups at 12 months. The secondary endpoints are relapse time, response rate and side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fulfillment of the 2019 American College of Rheumatology/European League against Rheumatology (ACR/EULAR) IgG4-related disease classification criteria; 2. Newly-onset or relapsed patients who requires initiation or continuation of glucocorticoids treatment; 3. The addition of glucocorticoids was started at lower than 10 mg/d.

Exclusion Criteria:

* 1. Patients who were diagnosed as other autoimmune diseases; 2. Patients who were diagnosed as malignant diseases; 3. Pregnant and lactating women； 4. Active infection: HIV, HCV, HBV, TB； 5. Severe irreversible damage of organ function; 6. Receipt of any biologic therapy or immunosuppressive agent other than GCs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The difference of relapse rate of IgG4-RD among 3 groups in 12 months. | 12 months
  The definition of relapse: elevation of IgG4-RD Responder Index ≥ 2 points; new organ involvement or recurrence, with or without elevation of serum IgG4 levels.

SECONDARY OUTCOMES:
The difference of the time at baseline to first relapse among 3 groups | 12 months
  The difference of The difference of relapse time in 3 groups
The difference of the response rate of the treatment among the 3 groups. | 12 months
  Complete response rate; Partial response rate; No response
Side effects | 12 months
  Any side effects caused by treatments for IgG4-RD.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China